CLINICAL TRIAL: NCT06736483
Title: Intravenous Dexmedetomidine as an Adjuvant to Locoregional Anesthesia in Pediatric Surgery: a Prospective, Randomized, Double-blind, Placebo-controlled Study. DEXPED
Brief Title: Intravenous Dexmedetomidine as an Adjuvant to Locoregional Anesthesia in Pediatric Surgery
Acronym: DEXPED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RECHMPL23_0433; 2024-514550-73-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia; Pediatric Surgery
Keywords: loco-regional anesthesia; Pain; Emergence delirium
MeSH Terms: conditions — Pain; Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Intravenous administration of 1 µg /kg of dexmedetomidine in 10 ml of 0.9% sodium chloride at the time of incision.
  Interventions: Drug: Dexmedetomidine; Other: Face Legs Activity Cry Consolability scale; Other: Post-Hospitalization Behavior Questionnaire; Other: Postoperative pain measure; Other: Post-operative quality of life questionnaire
- Placebo (Placebo Comparator): Intravenous administration of 10 ml sodium chloride 0.9% at the time of incision
  Interventions: Drug: Placebo administration; Other: Face Legs Activity Cry Consolability scale; Other: Post-Hospitalization Behavior Questionnaire; Other: Postoperative pain measure; Other: Post-operative quality of life questionnaire

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous administration of 1 µg /kg of dexmedetomidine in 10 ml of 0.9% sodium chloride at the time of incision.
  Arms: Dexmedetomidine
Drug: Placebo administration — Intravenous administration of 10 ml sodium chloride 0.9% at the time of incision
  Arms: Placebo
Other: Face Legs Activity Cry Consolability scale — The pain will be assessed on admission and every 15 minutes until discharge from the PACU
Other: Post-Hospitalization Behavior Questionnaire — The Post-Hospitalization Behavior Questionnaire will be completed at day 1 and at day 7
Other: Postoperative pain measure — The Postoperative pain measure will be completed by parents at day 1, day 7, 3 months and 6 months
Other: Post-operative quality of life questionnaire — The Post-operative quality of life questionnaire pedQL will be completed at 3 and 6 months

SUMMARY:
The main objective of this study is to study the impact of intravenous dexmedetomidine combined with locoregional anesthesia on postoperative pain in children undergoing surgery.

Secondary objectives was to compare beetwen groups : Post-operative pain; opioid consumption; incidence of emergence delirium, post-operative behavioral disorders, length of stay in the PACU, adverse events , parental satisfaction and quality of life.The goal of this clinical trial is to assess intravenous dexmedetomidine to prevent post-operative pain in children undergoing surgery.

This study is prospective and children will be randomized in one of the following arm:

* Dexmedetomidine (experimental treatment)
* Placebo The experimental treatment or placebo will be administrated at one time point at the time of incision.

Participants and their legal representative will have to respond to questionnaires at several time points following the surgery: Day 1, Week 1, Month 3 and Month 6.

DETAILED DESCRIPTION:
Postoperative pain, which can develop into chronic pain in children, can have a significant impact on the quality of life of the child and their parents. Management of acute postoperative pain is crucial to prevent chronic pain, and perioperative opioid sparing aims to reduce opioid side effects. The emergence of postoperative delirium (ED) is also a concern, as it can cause intense agitation and diagnostic difficulties. Dexmedetomidine, in addition to its sedative and analgesic effects, has been shown to prolong the duration and effectiveness of regional anesthesia (LAR), thereby reducing the need for opioids and attenuating the severity of postoperative delirium. Its use in these settings could improve pain management and reduce complications associated with pediatric surgery, thus offering a promising therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to 7 years old male or female
* To be hospitalized for scheduled urovisceral orchidopexy or peritoneovaginal canal surgery (inguinal hernia or hydrocele cure) on an outpatient basis
* Local-regional anesthesia via Transversus Abdominis Plane (TAP) block and/or pudendal block
* National health insurance coverage
* Have obtained signed informed consent from holders of parental authority
* American Society of Anesthesiology (ASA) score : 1-2
* French read, written and spoken by legal representatives

Exclusion Criteria:

* Patient under 1 or over 8 years old
* Patients with allergies to local anesthetics
* Patient with a contraindication to locoregional anesthesia: coagulation disorder or infection (fasciocutaneous) in the puncture zone
* Patients with a contraindication to dexmedetomidine (hypersensitivity to the active ingredient or one of the excipients, advanced heart block (level 2 or 3), uncontrolled hypotension, acute cerebrovascular pathologies)
* Patients with delayed psychological development, cognitive or behavioral disorders, or severe neurological pathology.
* Patients and/or parents who refused to participate in the study
* Proven allergy or contraindication to dexmedetomidine or nalbuphine
* Previous study participants

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-07-03 (Estimated); Study Completion 2028-07-03 (Estimated)

PRIMARY OUTCOMES:
Rescue analgesic | From the end of surgery to hospital discharge (up to 7 days)
  Rescue analgesic (Nalbuphine, Nubain®) administration in the PACU between the 2 arms.

SECONDARY OUTCOMES:
Postoperative pain | From the end of surgery to hospital discharge (up to 2 days)
  Assessment of postoperative pain using the Face Legs Activity Cry Consolability (FLACC) scale: on admission and every 15 minutes until discharge from the PACU, then before returning home.
Intraoperative morphine consumption | From anesthesia induction to the end of surgery (up to 24 hours)
Emergency analgesics | From the end of surgery to hospital discharge (up to 24 hours)
  Dose in milligrams of emergency analgesics in the PACU
Adverse events | From the end of surgery up to 7 postoperative days
  Incidence of opioid-related side effects (respiratory complications - postoperative nausea and vomiting)
Length of hospital stay | From the start of hospitalization to hospital discharge (up to 7 days)
  Length of hospital stay in hours from admission to discharge
Ped-PADSS score | From the end of surgery to hospital discharge (up to 2 days)
  The Post-Anesthetic Discharge Scoring System aimed to assess the possibility of discharge. The minimum is 0 and the maximum 10. A score of 9 or 10 authorizes hospital discharge.
Pediatric Anesthesia Emergence Delirium | From the end of surgery to hospital discharge (up to 24 hours)
  Incidence of emergence of delirium in the PACU according to the Pediatric Anesthesia Emergence Delirium (PAED) scale. Score from 0 to 20, a score > 9 indicates an emergence delirium
Post-Hospitalization Behavior Questionnaire | From the end of surgery up to 6 postoperative months
  Post-Hospitalization Behavior Questionnaire at day 1 and day 7. This questionnaire is composed of 27 items rated from 1 to 5, minimum score : 27, maximum score: 135. A score above 68 is associated with an increase in postoperative behavioral problems.
Postoperative Pain Measure For Parents | From the end of surgery up to 6 postoperative months
  Postoperative Pain Measure For Parents at 7 days, 3 and 6 months. Score: from 0 to 10 with 10 items. A score above 6 indicates significant pain.
Post-operative quality of life questionnaire | From the end of surgery up to 6 postoperative months
  Post-operative quality of life questionnaire pedsQL at 3 and 6 months. The 23 questions cover 4 different domains: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items).
  The parent questionnaire assesses parents' perceptions of their child's health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- UH of Montpellier, Montpellier, France, France